CLINICAL TRIAL: NCT05654818
Title: Peripheral Immunological Effects of High-dose Vitamin D Treatment in Healthy Subjects: Randomized, Single-center, Double-blind Trial
Brief Title: Peripheral Immunological Effects of High-dose Vitamin D Treatment in Healthy Subjects
Acronym: VDSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: CIVI/2021/ET-01; 2022-002157-25 (EudraCT Number)
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Vitamin d Deficiency
Keywords: Multiple sclerosis; Immunomodulation; lymphocyte subset
MeSH Terms: conditions — Vitamin D Deficiency; Multiple Sclerosis | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D (Experimental)
  Interventions: Drug: Vitamin D
- Control (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D — 100,000 UI
  Arms: Vitamin D
Drug: Placebo — The placebo is identical in appearance to the active treatment: a drinkable solution in ampoules that is clear, yellowish in color with a slightly lemony odor and an oily, slightly sweet, lemony taste.
  Arms: Control

SUMMARY:
Vitamin D deficiency is associated with the risk of developing MS. Vitamin D treatment has therefore been tested as a background treatment for this pathology, with a seemingly modest clinical effect. Indeed, the first therapeutic trials using high doses of vitamin D (SOLAR and CHOLINE) did not show a significant effect on short-term relapses. However, these two studies showed a significant decrease in the radiological activity of MS on MRI, suggesting a significant immunomodulatory efficacy but a weak clinical benefit in the short term.

Vitamin D has a pleiotropic effect on the immune system inducing overall immunomodulation through transcriptomic modulations, under the control of many individual genetic factors. However, in vivo, only one therapeutic trial has compared the immunological effect of Vitamin D in healthy subjects and in patients with a first demyelinating episode. Analysis of PBMC by flow cytometric cell sorting based on a very small number of markers (CD3, CD8, IL-17, IFN-g) did not find any significant quantitative modulation of Th17 or of their production of IL-10, IL-17 and IFN-g after treatment with Vitamin D measured by ELISA. However, the evolution of anti-inflammatory lymphocyte populations has not been evaluated. A few in vitro studies suggest that the effect of vitamin D may be incomplete on the lymphocytes of MS patients.

The study investigators will use an immunological FACS approach to describe activation markers and measure the intensity of changes induced in healthy subjects after 3 months of high-dose cholecalciferol versus placebo treatment using the same protocol as the D-Lay MS (NCT01817166) study.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* Women of childbearing potential must have effective contraception during the study period. Effective contraception is defined by a low failure rate (less than 1% per year) when used correctly and consistently, such as implants, injectables, oral contraceptives, IUDs, abstinence, or partner vasectomy. A urine pregnancy test will be performed at inclusion.

Exclusion Criteria:

* The subject is participating in another therapeutic study, or is in a period of exclusion determined by a previous study
* The subject is unable to express their consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* Pregnant or breastfeeding
* Infectious disease or vaccination within previous 3 months
* Chronic psychiatric disease, or disease that, in the opinion of the investigator ,may put the patient at risk or affect compliance.
* Chronic inflammatory or dysimmune disease or subject on immunomodulatory or immunosuppressive therapy (including corticosteroids) within the last 3 months.
* Uncontrolled epilepsy.
* Known vitamin D deficiency secondary to active or other digestive disease (celiac disease, IBD, gastrectomy or bypass, cirrhosis, short bowel syndrome, nephrotic syndrome, hyperthyroidism, hypoparathyroidism, cancer, granulomatous pathology, lymphoma, rickettsiosis).
* History of hypercalcemia, osteopenia or osteoporosis, urinary lithiasis, heart rhythm disorders.
* Pathology requiring a daily intake of more than 1 gram of Calcium.
* Contraindication to vitamin D3 treatment as mentioned on the VIDAL documentation of UVEDOSE.
* Treatment affecting vitamin D metabolism other than corticosteroids: anti-epileptic drugs [phenobarbital, primidone, phenytoin], rifampicin, isoniazid, ketoconazole, 5-FU and leucovorin, thiazide diuretic.
* Active vitamin supplementation or dietary supplements rich in vitamin D.
* Present or past neurological symptoms that may suggest an undiagnosed inflammatory neurological pathology.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2023-04-13 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Change in Lymphocyte T CD4+ cells since baseline | Month 3
  Percentage variation measured by Fluorescence Activated Cell Sorting of cells CD3+/CD4+
Change in T helper1 (Th1) Lymphocyte T CD4+ cells since baseline | Month 3
  Percentage variation measured by Fluorescence Activated Cell Sorting of cells CXCR3+ /CCR6-
Change in Th1*Lymphocyte T CD4+ cells since baseline | Month 3
  Percentage variation measured by Fluorescence Activated Cell Sorting of cells CXCR3+/CCR+
Change in naive Lymphocyte T CD4+ cells since baseline | Month 3
  Percentage variation measured by Fluorescence Activated Cell Sorting of cells CD45RA+/CCR7+
Change in effector memory Lymphocyte T CD4+ cells since baseline | Month 3
  Percentage variation measured by Fluorescence Activated Cell Sorting of cells CD45RA-/CCR7-
Change in central memory Lymphocyte T CD4+ cells since baseline | Month 3
  Percentage variation measured by Fluorescence Activated Cell Sorting of cells CD45RA-/CCR7+
Change in Teffector memory RA+ Lymphocyte T CD4+ cells since baseline | Month 3
  Percentage variation measured by Fluorescence Activated Cell Sorting of cells CD45RA+/CCR7-
Change in FOXP3 Treg / Treg Lymphocyte T CD4+ cells since baseline | Month 3
  Percentage variation measured by Fluorescence Activated Cell Sorting of cells CD25+/CD127+/FOXP3+
Change in naive Treg Lymphocyte T CD4+ cells since baseline | Month 3
  Percentage variation measured by Fluorescence Activated Cell Sorting of cells CD45RA+/FOXP3+
Change in memory Treg Lymphocyte T CD4+ cells since baseline | Month 3
  Percentage variation measured by Fluorescence Activated Cell Sorting of cells CD45RA-/FOXP3+
Change in Tr1 Lymphocyte T cells CD4+ since baseline | Month 3
  Percentage variation measured by Fluorescence Activated Cell Sorting of cells CD49b+/LAG3+
Change in Lymphocyte T CD8+ cells since baseline | Month 3
  Percentage variation measured by Fluorescence Activated Cell Sorting of cells CD3+/CD4-
Change in naive Lymphocyte T CD8+ cells since baseline | Month 3
  Percentage variation measured by Fluorescence Activated Cell Sorting of cells CD45RA+/CCR7+
Change in effector memory Lymphocyte T CD8+ cells since baseline | Month 3
  Percentage variation measured by Fluorescence Activated Cell Sorting of cells CD45RA-/CCR7-
Change in central memory Lymphocyte T CD8+ cells since baseline | Month 3
  Percentage variation measured by Fluorescence Activated Cell Sorting of cells CD45RA-/CCR7+
Change in Teffector memory RA+ Lymphocyte T CD8+ cells since baseline | Month 3
  Percentage variation measured by Fluorescence Activated Cell Sorting of cells CD45RA+/CCR7-
Change in Tc1 Lymphocyte T CD8+ cells since baseline | Month 3
  Percentage variation measured by Fluorescence Activated Cell Sorting of cells CXCR3+/CCR6-
Change in Tc1* Lymphocyte T CD8+ cells since baseline | Month 3
  Percentage variation measured by Fluorescence Activated Cell Sorting of cells CXCR3+/CCR6+
Change in Tc2 Lymphocyte T CD8+ cells since baseline | Month 3
  Percentage variation measured by Fluorescence Activated Cell Sorting of cells CXCR3-/CCR6-
Change in Tc17 Lymphocyte T CD8+ cells since baseline | Month 3
  Percentage variation measured by Fluorescence Activated Cell Sorting of cells CXCR3-/CCR6+
Change in CD8 Tcreg / TcReg Lymphocyte T CD8+ cells since baseline | Month 3
  Percentage variation measured by Fluorescence Activated Cell Sorting of cells CD25+/CD127+/FOXP3+
Change in naive Tcreg Lymphocyte T CD8+ cells since baseline | Month 3
  Percentage variation measured by Fluorescence Activated Cell Sorting of cells CD45RA+/FOXP3+
Change in memory Tcreg Lymphocyte T CD8+ cells since baseline | Month 3
  Percentage variation measured by Fluorescence Activated Cell Sorting of cells CD45RA-/FOXP3+
Change in Lymphocyte B cells since baseline | Month 3
  Percentage variation measured by Fluorescence Activated Cell Sorting of cells CD19+

SECONDARY OUTCOMES:
lymphocyte subpopulations change in CD6 phenotype after 3 months of high dose vitamin D treatment or placebo | Month 3
  Measured by Fluorescence Activated Cell Sorting of cells
lymphocyte subpopulations change in CD162 phenotype after 3 months of high dose vitamin D treatment or placebo | Month 3
  Measured by Fluorescence Activated Cell Sorting of cells
lymphocyte subpopulations change in CD226 phenotype after 3 months of high dose vitamin D treatment or placebo | Month 3
  Measured by Fluorescence Activated Cell Sorting of cells
lymphocyte subpopulations change in CD46 phenotype after 3 months of high dose vitamin D treatment or placebo | Month 3
  Measured by Fluorescence Activated Cell Sorting of cells
lymphocyte subpopulations change in CD11a phenotype after 3 months of high dose vitamin D treatment or placebo | Month 3
  Measured by Fluorescence Activated Cell Sorting of cells
lymphocyte subpopulations change in CD49d phenotype after 3 months of high dose vitamin D treatment or placebo | Month 3
  Measured by Fluorescence Activated Cell Sorting of cells
lymphocyte subpopulations change in CLA phenotype after 3 months of high dose vitamin D treatment or placebo | Month 3
  Measured by Fluorescence Activated Cell Sorting of cells
Change in production of cytokine IL-10 in lymphocyte subpopulations after 3 months of high dose vitamin D treatment or placebo | Month 3
  Measured by Fluorescence Activated Cell Sorting of cells
Change in production of cytokine IFNg in lymphocyte subpopulations after 3 months of high dose vitamin D treatment or placebo | Month 3
  Measured by Fluorescence Activated Cell Sorting of cells
Change in production of cytokine IL-17 in lymphocyte subpopulations after 3 months of high dose vitamin D treatment or placebo | Month 3
  Measured by Fluorescence Activated Cell Sorting of cells
Change in plasma Vitamin D levels 3 months after baseline of high dose Vitamin D treatment versus placebo | Month 3
  Determination of 25-OH-D2 and 25-OH-D3 forms in nmol/L in plasma with the "vitamin D total II" kit
Change in 16sRNA levels 3 months after baseline of high dose Vitamin D treatment versus placebo | Month 3
Nature of gut microbiota taxonomy 3 months after high dose Vitamin D treatment versus placebo | Month 3
  Number of operational taxonomic units
Nature of blood microbiota taxonomy 3 months after high dose Vitamin D treatment versus placebo | Month 3
  Number of operational taxonomic units
Percentage of gut microbiota taxonomy 3 months after high dose Vitamin D treatment versus placebo | Month 3
  Percentage of operational taxonomic units
Percentage of blood microbiota taxonomy 3 months after high dose Vitamin D treatment versus placebo | Month 3
  Percentage of operational taxonomic units
Diversity of gut microbiota 3 months after high dose Vitamin D treatment versus placebo | Month 3
  Shannon index
Diversity of blood microbiota 3 months after high dose Vitamin D treatment versus placebo | Month 3
  Shannon index
Beta diversity of gut microbiota 3 months after high dose Vitamin D treatment versus placebo | Month 3
  Bray-Curtis index
Beta diversity of blood microbiota 3 months after high dose Vitamin D treatment versus placebo | Month 3
  Bray-Curtis index
Describing the genetic determinants of vitamin D response using a Single Nucleotide Polymorphism (SNP) database | Month 3
  Description of individual SNPs

CONTACTS AND LOCATIONS:
Overall Officials: Eric Thouvenot, Principal Investigator — CHU de Nimes
Locations (1):
- CHU de Nîmes, Nîmes, France